CLINICAL TRIAL: NCT02795585
Title: Feasibility of On-line Computed Fractional Flow Reserve: The Wire-free Invasive Functional Imaging (WIFI) Study
Brief Title: The Wire-free Invasive Functional Imaging (WIFI) Study
Acronym: WIFI
Status: Completed | Type: Observational
Sponsor: Niels Ramsing Holm (Other)
Responsible Party: Sponsor-Investigator, Niels Ramsing Holm, Research associate, M.D., Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Other Study IDs: 1-10-72-272-15
Record Dates: First submitted 2016-04-29; First posted 2016-06-10 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Coronary Artery Disease
Keywords: Fractional Flow Reserve; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- QFR group: Patients with stable angina pectoris and indication for FFR.
  Interventions: Other: QFR (observational)

INTERVENTIONS:
Other: QFR (observational) — QFR assessment by Medis Suite, Medis medical imaging B.V., The Netherlands

SUMMARY:
Quantitative Flow Ratio (QFR) is a new method for evaluating the functional significance of coronary stenosis by calculation of the pressure in the vessel based on two angiographic projections. The purpose of the WIFI study is to evaluate feasibility of QFR when performed during coronary angiography and compare diagnostic accuracy to standard FFR.

DETAILED DESCRIPTION:
Background:

Patients at high risk of having one or more coronary stenosis are evaluated routinely by invasive coronary angiography (CAG) and often in combination with measurement of fractional flow reserve (FFR) to assess the functional significance of identified stenosis. FFR is assessed during CAG by advancing a wire with a pressure transducer towards the stenosis and measure the ratio in pressure between the two sides of the stenosis during maximum blood flow (hyperaemia) induced by adenosine infusion.

The solid evidence for FFR evaluation of coronary stenosis and the relative simplicity in performing the measurements have supported adoption of an FFR based strategy in many centers but the need for interrogating the stenosis by a pressure wire and the cost of the wire and the drug inducing hyperaemia limits more widespread adoption.

Quantitative Flow Ratio is a novel method for evaluating the functional significance of coronary stenosis by calculation of the pressure in the vessel based on two angiographic projections.

The purpose of the WIFI study is to evaluate feasibility of QFR when performed during coronary angiography and compare diagnostic accuracy to standard FFR.

Hypothesis:

QFR can be assessed during CAG for stenosis interrogated by FFR

Methods:

Proof-of-concept, prospective, observational, single arm study with inclusion of 100 patients. Clinical follow-up by telephone call after one year.

A stenosis with indication for FFR is identified and at least two angiographic projections rotated at least 25 degrees around the target vessel are acquired during resting conditions. QFR is calculated on-line using the Medis Suite application and simultaneously to the operator performing the FFR measurement using I.V. adenosine. The QFR observer is blinded to the FFR measurement.

QFR is reassessed off-line by internal observer and by an external core laboratory. Both blinded to FFR results.

FFR is assessed in core laboratory by a different blinded observer

All data are entered and stored in a protected and logged trial management system (TrialPartner).

ELIGIBILITY:
Inclusion Criteria:

* Stable angina pectoris and secondary evaluation of stenosis after acute myocardial infarction (AMI)
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* Myocardial infarction within 72 hours
* Severe asthma and chronic obstructive pulmonary disease
* Severe heart failure (NYHA≥III)
* S-creatinine>120µmol/L
* Allergy to contrast media or adenosine
* Stenosis in vein graft
* Ostial left main stenosis
* Severe tortuosity
* Atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable angina pectoris admitted for coronary angiography due to high risk of significant coronary stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2016-06-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of in-procedure QFR | 1 hour
  Percentage of successful QFR in FFR-cases.

SECONDARY OUTCOMES:
Proportion of patients with positive QFR of FFR positive patients (true positives) (sensitivity) | 1 hour
  Positive FFR is defined as FFR≤0.80. Positive QFR is defined as QFR≤0.80
Proportion of patients with negative QFR of patients with negative FFR (true negatives) (specificity) | 1 hour
  Negative FFR is defined as FFR>0.80. Negative QFR is defined as QFR>0.80
Proportion of patients with positive FFR (true positives) of patients with positive QFR (positive predictive value) | 1 hour
  Positive FFR is defined as FFR≤0.80. Positive QFR is defined as QFR≤0.80
Proportion of patients with negative FFR (true negatives) of patients with negative QFR (negative predictive value) | 1 hour
  Negative FFR is defined as FFR>0.80. Negative QFR is defined as QFR>0.80
Diagnostic performance of QFR in comparison to FFR reported as positive and negative likelihood ratio | 1 hour
Diagnostic accuracy of QFR in comparison to 2D quantitative coronary angiography (QCA) (>50% diameter stenosis) | 1 hour
  Defined as area under the receiver operating curve (ROC)
Diagnostic accuracy of QFR based on fixed hyperemic flow rate (in-procedure analysis) | 1 hour
  Defined as area under the receiver operating curve (ROC)
Diagnostic accuracy of QFR based on Thrombolysis in Myocardial Infarction(TIMI) flow without hyperemia (in-procedure analysis) | 1 hour
  Defined as area under the receiver operating curve (ROC)
Diagnostic accuracy of QFR based on TIMI flow with hyperemia (core laboratory analysis) | 1 hour
  Defined as area under the receiver operating curve (ROC)
Any QFR procedure-related adverse events/complications (safety) | 1 hour
  Death, myocardial infarction, acute renal failure clearly related to additional angiographic projections.
Time to FFR | 1 hour
  From last diagnostic angiogram before advancing FFR-wire to approved drift-check
Time to QFR | 1 hour
  From receiving angiographic images to QFR-value
Contrast use | 1 hour
  Volume of contrast for total procedure
Fluoroscopy time | 1 hour
Myocardial infarction | 1 year
  Universal definition
Target lesion failure | 1 year
  Universal definition
Target lesion revascularization | 1 year
  Universal definition
Stent thrombosis | 1 year
  Universal definition
Angina pectoris | 1 year
  Canadian Cardiovascular Society (CCS)-class
Cardiac death | 1 year
  Universal definition
Non-cardiac death | 1 year
  Universal definition

CONTACTS AND LOCATIONS:
Overall Officials: Niels R. Holm, M.D., Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hspital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided